CLINICAL TRIAL: NCT01047501
Title: Evaluation of the Effect of Two Doses of AMR101 (Ethyl Icosapentate) on Fasting Serum Triglyceride Levels in Patients With Persistent High Triglyceride Levels (≥ 200 mg/dL and < 500 mg/dL) Despite Statin Therapy
Brief Title: Effect of AMR101 (Ethyl Icosapentate) on Triglyceride (Tg) Levels in Patients on Statins With High Tg Levels (≥ 200 and < 500 mg/dL)
Acronym: ANCHOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amarin Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMR-01-01-0017; The ANCHOR Study (Other: Amarin Pharma Inc.)
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Hypertriglyceridemia
Keywords: hypertriglyceridemia; omega-3 fatty acids; statin; triglycerides; lipids; EPA; docosahexaenoic acid; fish; fatty acids; fibrates; niacin; lipid; atorvastatin; Lovaza; simvastatin; lovastatin; pravastatin; fluvastatin; rosuvastatin; Trilipix; Vytorin; Simcor; Niaspan; ezetimibe; Zetia; ethyl-EPA; ethyl icosapentate; Crestor; Zocor; Lipitor; LDL; HDL; cholesterol; dyslipidemia; VASCEPA; icosapent ethyl
MeSH Terms: conditions — Hypertriglyceridemia; Dyslipidemias | interventions — eicosapentaenoic acid ethyl ester; eicosapentaenoic acid ethanolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- AMR101 (ethyl icosapentate) - 2 g/day (Experimental)
  Interventions: Drug: AMR101 (ethyl icosapentate) - 2 g/day
- AMR101 (ethyl icosapentate) - 4 g/day (Experimental)
  Interventions: Drug: AMR101 (ethyl icosapentate) - 4 g/day

INTERVENTIONS:
Drug: AMR101 (ethyl icosapentate) - 4 g/day — AMR101 (ethyl icosapentate) 4 capsules/day for 12 weeks
  Other Names: VASCEPA® (icosapent ethyl)
  Arms: AMR101 (ethyl icosapentate) - 4 g/day
Drug: AMR101 (ethyl icosapentate) - 2 g/day — AMR101 (ethyl icosapentate) 2 capsules/day with placebo 2 capsules/day for 12 weeks
  Other Names: VASCEPA® (icosapent ethyl)
  Arms: AMR101 (ethyl icosapentate) - 2 g/day
Drug: Placebo — Placebo 4 capsules/day for 12 weeks
  Arms: Placebo

SUMMARY:
The primary objective is to determine the efficacy of AMR101 (ethyl icosapentate) compared to placebo in lowering high fasting triglyceride levels in patients with high risk for cardiovascular disease and fasting triglyceride levels ≥ 200 and < 500 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages >18
* Fasting triglyceride ≥200 mg/dL and <500 mg/dL
* LDL-C (low density lipoprotein - cholesterol) ≥40 mg/dL and <100 mg/dL
* High risk for coronary heart disease
* On stable dose of statin (atorvastatin, rosuvastatin or simvastatin)
* Provide written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant
* Use of non-statin lipid-altering drugs which cannot be stopped including fibrates, niacin, fish oil and other products containing omega-3 fatty acids or other dietary supplements with potential lipid-altering effects
* History of bariatric surgery or currently on weight loss drugs
* Uncontrolled hypertension (BP > 160/100)
* HIV infection or on treatment with HIV-protease inhibitors, cyclophosphamide,or isotretinoin
* Consumption of more than 2 alcoholic beverages per day
* History of cancers (except if been disease free for >5 years OR history was basal or squamous cell skin cancer)
* Participation in another clinical trial involving an investigational agent in the last 30 days
* Other parameters will be assessed at the study center to ensure eligibility for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (72):
  - Amarin Investigational Site, Muscle Shoals, Alabama
  - Amarin Investigational Site, Scottsboro, Alabama
  - Amarin Investigational Site, Phoenix, Arizona
  - Amarin Investigational Site, Tucson, Arizona
  - Amarin Investigational Site, Anaheim, California
  - Amarin Investigational Site, Burbank, California
  - Amarin Investigational Site, Chino, California
  - Amarin Investigational Site, Encinitas, California
  - Amarin Investigational Site, Irvine, California
  - Amarin Investigational Site, Los Angeles, California
  - Amarin Investigational Site, Spring Valley, California
  - Amarin Investigational Site, Westlake Village, California
  - Amarin Investigational Site, Golden, Colorado
  - Amarin Investigational Site, Wheat Ridge, Colorado
  - Amarin Investigational Site, Aventura, Florida
  - Amarin Investigational Site, Clearwater, Florida
  - Amarin Investigational Site, Coral Gables, Florida
  - Amarin Investigational Site, Hialeah, Florida
  - Amarin Investigational Site, Jacksonville, Florida
  - Amarin Investigational Site, Miami, Florida
  - Amarin Investigational Site, New Port Richey, Florida
  - Amarin Investigational Site, Orlando, Florida
  - Amarin Investigational Site, Port Orange, Florida
  - Amarin Investigational Site, West Palm Beach, Florida
  - Amarin Investigational Site, Augusta, Georgia
  - Amarin Investigational Site, Addison, Illinois
  - Amarin Investigational Site, Morton, Illinois
  - Amarin Investigational Site, Indianapolis, Indiana
  - Amarin Investigational Site, Kansas City, Kansas
  - Amarin Investigational Site, Newton, Kansas
  - Amarin Investigational Site, Wichita, Kansas
  - Amarin Investigational Site, Louisville, Kentucky
  - Amarin Investigational Site, Munfordville, Kentucky
  - Amarin Investigational Site, Auburn, Maine
  - Amarin Investigational Site, Baltimore, Maryland
  - Amarin Investigational Site, Elkridge, Maryland
  - Amarin Investigational Site, Troy, Michigan
  - Amarin Investigational Site, Olive Branch, Mississippi
  - Amarin Investigational Site, St Louis, Missouri
  - Amarin Investigational Site, Butte, Montana
  - Amarin Investigational Site, Concord, New Hampshire
  - Amarin Investigational Site, Endwell, New York
  - Amarin Investigational Site, New Windsor, New York
  - Amarin Investigational Site, Syracuse, New York
  - Amarin Investigational Site, Charlotte, North Carolina
  - Amarin Investigational Site, Durham, North Carolina
  - Amarin Investigational Site, Hickory, North Carolina
  - Amarin Investigational Site, Raleigh, North Carolina
  - Amarin Investigational Site, Statesville, North Carolina
  - Amarin Investigational Site, Wilmington, North Carolina
  - Amarin Investigational Site, Winston-Salem, North Carolina
  - Amarin Investigational Site, Cincinnati, Ohio
  - Amarin Investigational Site, Cleveland, Ohio
  - Amarin Investigational Site, Kettering, Ohio
  - Amarin Investigational Site, Norman, Oklahoma
  - Amarin Investigational Site, Tulsa, Oklahoma
  - Amarin Investigational Site, Beaver, Pennsylvania
  - Amarin Investigational Site, Harleysville, Pennsylvania
  - Amarin Investigational Site, Jersey Shore, Pennsylvania
  - Amarin Investigational Site, Lansdale, Pennsylvania
  - Amarin Investigational Site, Philadelphia, Pennsylvania
  - Amarin Investigational Site, Mt. Pleasant, South Carolina
  - Amarin Investigational Site, Rapid City, South Dakota
  - Amarin Investigational Site, Dallas, Texas
  - Amarin Investigational Site, Houston, Texas
  - Amarin Investigational Site, Lake Jackson, Texas
  - Amarin Investigational Site, San Antonio, Texas
  - Amarin Investigational Site, Temple, Texas
  - Amarin Investigational Site, Ettrick, Virginia
  - Amarin Investigational Site, Norfolk, Virginia
  - Amarin Investigational Site, Richmond, Virginia
  - Amarin Investigational Site, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ballantyne CM, Bays HE, Kastelein JJ, Stein E, Isaacsohn JL, Braeckman RA, Soni PN. Efficacy and safety of eicosapentaenoic acid ethyl ester (AMR101) therapy in statin-treated patients with persistent high triglycerides (from the ANCHOR study). Am J Cardiol. 2012 Oct 1;110(7):984-92. doi: 10.1016/j.amjcard.2012.05.031. Epub 2012 Jul 20. PMID 22819432
- [Result] Brinton EA, Ballantyne CM, Bays HE, Kastelein JJ, Braeckman RA, Soni PN. Effects of icosapent ethyl on lipid and inflammatory parameters in patients with diabetes mellitus-2, residual elevated triglycerides (200-500 mg/dL), and on statin therapy at LDL-C goal: the ANCHOR study. Cardiovasc Diabetol. 2013 Jul 9;12:100. doi: 10.1186/1475-2840-12-100. PMID 23835245
- [Result] Bays HE, Ballantyne CM, Braeckman RA, Stirtan WG, Soni PN. Icosapent ethyl, a pure ethyl ester of eicosapentaenoic acid: effects on circulating markers of inflammation from the MARINE and ANCHOR studies. Am J Cardiovasc Drugs. 2013 Feb;13(1):37-46. doi: 10.1007/s40256-012-0002-3. PMID 23325450
- [Result] Ballantyne CM, Braeckman RA, Bays HE, Kastelein JJ, Otvos JD, Stirtan WG, Doyle RT Jr, Soni PN, Juliano RA. Effects of icosapent ethyl on lipoprotein particle concentration and size in statin-treated patients with persistent high triglycerides (the ANCHOR Study). J Clin Lipidol. 2015 May-Jun;9(3):377-83. doi: 10.1016/j.jacl.2014.11.009. Epub 2014 Nov 29. PMID 26073397
- [Result] Bays HE, Ballantyne CM, Braeckman RA, Stirtan WG, Doyle RT Jr, Philip S, Soni PN, Juliano RA. Icosapent Ethyl (Eicosapentaenoic Acid Ethyl Ester): Effects Upon High-Sensitivity C-Reactive Protein and Lipid Parameters in Patients With Metabolic Syndrome. Metab Syndr Relat Disord. 2015 Aug;13(6):239-47. doi: 10.1089/met.2014.0137. Epub 2015 Apr 20. PMID 25893544
- [Result] Ballantyne CM, Bays HE, Braeckman RA, Philip S, Stirtan WG, Doyle RT Jr, Soni PN, Juliano RA. Icosapent ethyl (eicosapentaenoic acid ethyl ester): Effects on plasma apolipoprotein C-III levels in patients from the MARINE and ANCHOR studies. J Clin Lipidol. 2016 May-Jun;10(3):635-645.e1. doi: 10.1016/j.jacl.2016.02.008. Epub 2016 Feb 23. PMID 27206952
- [Result] Ballantyne CM, Bays HE, Philip S, Doyle RT Jr, Braeckman RA, Stirtan WG, Soni PN, Juliano RA. Icosapent ethyl (eicosapentaenoic acid ethyl ester): Effects on remnant-like particle cholesterol from the MARINE and ANCHOR studies. Atherosclerosis. 2016 Oct;253:81-87. doi: 10.1016/j.atherosclerosis.2016.08.005. Epub 2016 Aug 20. PMID 27596132
- [Result] Bays HE, Ballantyne CM, Doyle RT Jr, Juliano RA, Philip S. Icosapent ethyl: Eicosapentaenoic acid concentration and triglyceride-lowering effects across clinical studies. Prostaglandins Other Lipid Mediat. 2016 Sep;125:57-64. doi: 10.1016/j.prostaglandins.2016.07.007. Epub 2016 Jul 11. PMID 27418543
- [Result] Mosca L, Ballantyne CM, Bays HE, Guyton JR, Philip S, Doyle RT Jr, Juliano RA. Usefulness of Icosapent Ethyl (Eicosapentaenoic Acid Ethyl Ester) in Women to Lower Triglyceride Levels (Results from the MARINE and ANCHOR Trials). Am J Cardiol. 2017 Feb 1;119(3):397-403. doi: 10.1016/j.amjcard.2016.10.027. Epub 2016 Nov 1. PMID 27939227
- [Result] Brinton EA, Ballantyne CM, Guyton JR, Philip S, Doyle RT Jr, Juliano RA, Mosca L. Lipid Effects of Icosapent Ethyl in Women with Diabetes Mellitus and Persistent High Triglycerides on Statin Treatment: ANCHOR Trial Subanalysis. J Womens Health (Larchmt). 2018 Sep;27(9):1170-1176. doi: 10.1089/jwh.2017.6757. Epub 2018 Mar 27. PMID 29583081
- [Result] Miller M, Ballantyne CM, Bays HE, Granowitz C, Doyle RT Jr, Juliano RA, Philip S. Effects of Icosapent Ethyl (Eicosapentaenoic Acid Ethyl Ester) on Atherogenic Lipid/Lipoprotein, Apolipoprotein, and Inflammatory Parameters in Patients With Elevated High-Sensitivity C-Reactive Protein (from the ANCHOR Study). Am J Cardiol. 2019 Sep 1;124(5):696-701. doi: 10.1016/j.amjcard.2019.05.057. Epub 2019 Jun 6. PMID 31277790
- [Result] Ballantyne CM, Manku MS, Bays HE, Philip S, Granowitz C, Doyle RT Jr, Juliano RA. Icosapent Ethyl Effects on Fatty Acid Profiles in Statin-Treated Patients With High Triglycerides: The Randomized, Placebo-controlled ANCHOR Study. Cardiol Ther. 2019 Jun;8(1):79-90. doi: 10.1007/s40119-019-0131-8. Epub 2019 Feb 20. PMID 30788718
- [Result] Vijayaraghavan K, Szerlip HM, Ballantyne CM, Bays HE, Philip S, Doyle RT Jr, Juliano RA, Granowitz C. Icosapent ethyl reduces atherogenic markers in high-risk statin-treated patients with stage 3 chronic kidney disease and high triglycerides. Postgrad Med. 2019 Aug;131(6):390-396. doi: 10.1080/00325481.2019.1643633. Epub 2019 Jul 25. PMID 31306043

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day
Started | 233 | 236 | 233
Completed | 217 | 225 | 221
Not Completed | 16 | 11 | 12
Not completed — Adverse Event | 7 | 8 | 5
Not completed — Withdrew Consent | 6 | 2 | 4
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Triglycerides >800 mg/dL | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Other discontinuation | 1 | 0 | 1
Not completed — Investigator judgement | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Total
Number analyzed (Participants) | 233 | 236 | 233 | 702
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.05) | 61.8 (9.42) | 61.1 (10.03) | 61.4 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 92 | 91 | 271
  Male | 145 | 144 | 142 | 431
Race/Ethnicity, Customized [Number; unit: participants]
  White | 224 | 226 | 226 | 676
  Other | 9 | 10 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Triglyceride Lowering Effect
Description: Median percent change from baseline to Week 12 in fasting serum triglyceride levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: Intent-to-treat population: randomized patients who received >= 1 dose of study drug and had baseline and >= 1 postrandomization efficacy measurement. Only patients with non-missing baseline and Week 12 endpoint values were included.
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 234 | 226 | 227
Percent change from baseline | -5.6 [-21.1 to 13.4] | -17.5 [-30.5 to 0.5] | 5.9 [-13.5 to 31.3]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; A sample size of 194 was required to provide 90.6% power to detect a difference of 15% between AMR101 4 g/day and placebo in percent change from baseline in fasting TG levels, assuming an SD of 45% in TG measurements and a significance level (p value) of 0.05, and 80% power to demonstrate noninferiority (p 0.025, 1-sided) of the LDL-cholesterol response between AMR101 4 g/day and placebo with a +6% margin. To accommodate a 10% drop-out rate, recruitment was planned for 648 randomized patients; Test type: Superiority or Other; p < 0.0001, Wilcoxon rank-sum test — Nonparametric analysis p values were planned using Wilcoxon rank-sum test for each comparison between AMR101 and placebo. Comparisons between AMR101 and placebo were made using a significance level of 0.05; A prespecified step-down testing procedure was used to control Type I error rate using 4 g/day vs placebo then, if significant, 2 g/day vs placebo; Median Difference (Final Values) = -21.5, 95% CI 2-sided [-26.7 to -16.2] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0005, Wilcoxon rank-sum test; Median Difference (Final Values) = -10.1, 95% CI 2-sided [-15.7 to -4.5] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

2. Secondary Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Low-density Lipoprotein Cholesterol Levels
Description: Median percent change from baseline to Week 12 in serum low density lipoprotein cholesterol levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 233 | 225 | 226
Percent change from baseline | 2.4 [-8.3 to 17.7] | 1.5 [-11.6 to 15.0] | 8.8 [-7.8 to 23.2]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Nonparametric analysis p values were planned using Wilcoxon rank-sum test for each comparison between AMR101 and placebo with a significance level of 0.05. Non-inferiority tests for percent change from baseline in LDL-C were performed between AMR101 and placebo to determine if AMR101 was statistically non-inferior to placebo with regard to increases in LDL-C. The pre-specified LDL-C criterion for noninferiority was the upper boundary 97.5% confidence interval not crossing the +6% threshold; p = 0.0067, Wilcoxon rank-sum test; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -6.2, 95% CI 2-sided [-10.5 to -1.7] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.0867, Wilcoxon rank-sum test; Median Difference (Final Values) = -3.6, 95% CI 2-sided [-7.9 to 0.5] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

3. Secondary Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Non-High-Density Lipoprotein Cholesterol Levels
Description: Median percent change from baseline to Week 12 in serum non-high density lipoprotein cholesterol levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 234 | 226 | 227
Percent change from baseline | 2.4 [-7.0 to 19.0] | -5.0 [-13.5 to 7.8] | 9.8 [-3.5 to 24.1]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -13.6, 95% CI 2-sided [-17.2 to -9.9] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0140, Wilcoxon rank-sum test; Median Difference (Final Values) = -5.5, 95% CI 2-sided [-9.4 to -1.7] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

4. Secondary Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Very Low-density Lipoprotein Cholesterol Levels
Description: Median percent change from baseline to Week 12 in serum very low-density lipoprotein cholesterol levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 233 | 225 | 226
Percent change from baseline | 1.6 [-20.0 to 34.5] | -12.1 [-31.3 to 16.7] | 15.0 [-10.9 to 47.8]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -24.4, 95% CI 2-sided [-31.9 to -17.0] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0170, Wilcoxon rank-sum test; Median Difference (Final Values) = -10.5, 95% CI 2-sided [-18.3 to -2.5] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

5. Secondary Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Lipoprotein-associated Phospholipase A2 Levels
Description: Median percent change from baseline to Week 12 in serum Lipoprotein-associated Phospholipase A2 levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 224 | 217 | 213
Percent change from baseline | -1.8 [-12.7 to 10.4] | -12.8 [-22.1 to -3.6] | 6.7 [-6.4 to 17.6]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -19.0, 95% CI 2-sided [-22.2 to -15.7] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0004, Wilcoxon rank-sum test; Median Difference (Final Values) = -8.0, 95% CI 2-sided [-11.6 to -4.5] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

6. Secondary Outcome: Difference Between AMR101 (Ethyl Icosapentate) and Placebo Treatment Groups in Apolipoprotein B Levels
Description: Median percent change from baseline to Week 12 in serum Apolipoprotein B levels following treatment with AMR101 (ethyl icosapentate) 2 g/day or 4 g/day
Time Frame: baseline and 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change from baseline
Arm/Group | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day | Placebo
Number analyzed (Participants) | 227 | 217 | 219
Percent change from baseline | 1.6 [-6.4 to 14.3] | -2.2 [-10.2 to 6.2] | 7.1 [-4.7 to 18.6]
Statistical Analysis 1: Comparison: AMR101 (Ethyl Icosapentate) - 4 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0001, Wilcoxon rank-sum test — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -9.3, 95% CI 2-sided [-12.3 to -6.1] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method
Statistical Analysis 2: Comparison: AMR101 (Ethyl Icosapentate) - 2 g/Day vs Placebo; Test type: Superiority or Other; p = 0.0170, Wilcoxon rank-sum test; Median Difference (Final Values) = -3.8, 95% CI 2-sided [-6.9 to -0.7] — Median differences between the treatment groups and 95% CIs were estimated with the Hodges-Lehmann method

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Events were collected by systematic assessment at each study visit.
Arm/Group | Placebo | AMR101 (Ethyl Icosapentate) - 2 g/Day | AMR101 (Ethyl Icosapentate) - 4 g/Day
Serious Adverse Events (participants affected / at risk) | 5/233 | 6/236 | 7/233
Other Adverse Events (participants affected / at risk) | 25/233 | 28/236 | 18/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=233) | AMR101 (Ethyl Icosapentate) - 2 g/Day (N=236) | AMR101 (Ethyl Icosapentate) - 4 g/Day (N=233)
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Angina, unstable (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=233) | AMR101 (Ethyl Icosapentate) - 2 g/Day (N=236) | AMR101 (Ethyl Icosapentate) - 4 g/Day (N=233)
Diarrhea (Gastrointestinal disorders) | 10 | 9 | 8
Nasopharyngitis (Infections and infestations) | 7 | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 8 | 4
Nausea (Gastrointestinal disorders) | 7 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs are restricted in sharing data until an abstract presentation or publication of the manuscript.